CLINICAL TRIAL: NCT06029335
Title: Clinical Risk Assessment of Cognitive Function in Systemic Autoimmune Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, dr Varjú Cecília, Associate Professor, University of Pecs
Other Study IDs: 35147-3/2020/ EÜIG; 05570-6/2023 (Other: National Public Health Centre Institutional Committee of Science and Research Ethics Hungary)
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Systemic Sclerosis; Systemic Lupus Erythematosus; Myopathies, Inflammatory; Rheumatoid Arthritis; Healthy
MeSH Terms: conditions — Scleroderma, Systemic; Lupus Erythematosus, Systemic; Myositis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Investigations of serum samples for biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Diffuse cutaneous Systemic sclerosis: Physical examination, routine blood, immunoserology, and special biomarker laboratory examination. General health, functional, and quality of life questionnaires, and neuropsychological measures are administered.
- Limited cutaneous Systemic sclerosis: Physical examination, routine blood, immunoserology, and special biomarker laboratory examination. General health, functional, and quality of life questionnaires, and neuropsychological measures are administered.
- Primary Raynaud's: Physical examination, routine blood, immunoserology, and special biomarker laboratory examination. General health, functional, and quality of life questionnaires, and neuropsychological measures are administered.
- Healthy: Physical examination, routine blood, immunoserology, and special biomarker laboratory examination. General health, functional, and quality of life questionnaires, and neuropsychological measures are administered.
- Rheumatoid arthritis: Physical examination, routine blood, immunoserology, and special biomarker laboratory examination. General health, functional, and quality of life questionnaires, and neuropsychological measures are administered.
- Inflammatory myopathies: Physical examination, routine blood, immunoserology, and special biomarker laboratory examination. General health, functional, and quality of life questionnaires, and neuropsychological measures are administered.
- Systemic lupus erythematosus: Physical examination, routine blood, immunoserology, and special biomarker laboratory examination. General health, functional, and quality of life questionnaires, and neuropsychological measures are administered.

SUMMARY:
Objectives: Systemic autoimmune diseases are chronic diseases characterized by chronic inflammation, vasculopathy, and autoimmune phenomena. Several organ involvements are typical, including the central nervous system. Formerly published investigations emphasize a mild cognitive impairment affecting attention, memory, and complicated solution tasks. However, these symptoms significantly impact patients' routines and quality of life. The study examined the associations between cognitive impairment and clinical parameters regarding systemic autoimmune diseases.

Methods: General clinical data, some serum biomarkers including CCl-18, YKL-40, COMP, VEGF, Galectin-3, and Pentraxin as well as results of functional, quality of life, and neuropsychological measures, the Mini-Mental State Examination (MMSE), the Digit Span Forward-Backward, the Trail making A, B and the Digit Symbol tests all were administered.

ELIGIBILITY:
Inclusion Criteria:

* Systemic autoimmune diseases
* Healthy individuals - as controls

Exclusion Criteria:

* Diseases of the central nervous system
* Presence of pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients were enrolled into the study originating from the Rheumatology and Immunology Department, Medical School, University of Pécs.
  Control healthy groups including consecutive sex and age-matched healthy individuals are invited to participate.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Mini-mental State Examination | 12 months
  Complex Cognitive measure
The Functional Assessment of Chronic Illness Therapy F | 12 months
  health-related quality of life measure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pécs, Department of Rheumatology and Immunology, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No
Data are not publicly available due to ethical issues.

REFERENCES:
- [Background] Olah C, Schwartz N, Denton C, Kardos Z, Putterman C, Szekanecz Z. Cognitive dysfunction in autoimmune rheumatic diseases. Arthritis Res Ther. 2020 Apr 15;22(1):78. doi: 10.1186/s13075-020-02180-5. PMID 32293528
- [Derived] Krampek L, Kiss F, Farkas N, Faludi R, Nagy G, Szabo A, Czirjak L, Varju C. Risk factors of cognitive function impairment in patients with systemic sclerosis. Clin Exp Rheumatol. 2025 Aug;43(8):1481-1491. doi: 10.55563/clinexprheumatol/isx6h8. Epub 2025 Aug 1. PMID 40757427